CLINICAL TRIAL: NCT04422951
Title: Wise Social Psychological Interventions to Improve Outcomes of Behavioral Weight Control in Children With Obesity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Delays and complications due to the Covid pandemic
Sponsor: Stanford University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Thomas Robinson, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 54341; R01DK123286 (NIH)
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Results first posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity | interventions — Educational Status

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wise interventions plus behavioral Rx (Experimental): Wise social psychological interventions (growth mindset and values self-affirmation) plus a usual care behavioral intervention for weight control.
  Interventions: Behavioral: Wise interventions -- values self-affirmation and growth mindset -- plus usual care behavioral treatment
- Education plus behavioral Rx (Active Comparator): Health education plus a usual care behavioral intervention for weight control
  Interventions: Behavioral: Education plus usual care behavioral treatment

INTERVENTIONS:
Behavioral: Wise interventions -- values self-affirmation and growth mindset -- plus usual care behavioral treatment — Addition of two wise wise social psychological interventions-growth mindset and self-affirmation-to a 6-month usual care behavioral intervention for weight control in children with obesity
  Arms: Wise interventions plus behavioral Rx
Behavioral: Education plus usual care behavioral treatment — 6-month health education plus usual care behavioral intervention for weight control in children with obesity
  Arms: Education plus behavioral Rx

SUMMARY:
A 2-arm, parallel group, randomized controlled trial to evaluate overall differences in body mass index (BMI) trajectories over 6 months between 10-16-year-old children with obesity randomized to receive the wise social psychological interventions plus a usual care behavioral intervention for weight management compared to children randomized to receive additional education plus a usual care behavioral intervention.

ELIGIBILITY:
Inclusion Criteria:

* 10-16 year old children with obesity (BMI ≥ 95th percentile on the 2000 Centers for Disease Control and Prevention BMI reference) on the date of randomization. Participation in a behavioral weight control program. Standard behavioral weight control program eligibility criteria will apply: Child and at least one parent/guardian must agree to participate

Exclusion Criteria:

* Medical conditions affecting growth - diagnosed with a genetic or metabolic disease/syndrome associated obesity, Type 1 diabetes, Type 2 diabetes taking medication, chronic gastrointestinal diseases, Chronic renal diseases, uncorrected structural heart disease, heart failure, heart transplant, anorexia nervosa or bulimia nervosa or binge eating disorder (present or past), AIDS or HIV infection, pregnancy

Medications affecting growth - systemic corticosteroids more than 2 weeks in the past year, insulin, oral hypoglycemics, thyroid hormone, growth hormone

Conditions limiting participation in the interventions - e.g., unable to participate in routine physical education classes at school, requiring oxygen supplementation for exertion, developmental or physical disability preventing participation in interventions, children or parents/guardians who cannot medically participate in mild dietary restrictions and/or increased physical activity for any reason

Conditions limiting participation in the assessments - child or primary caregiver not able to read surveys in English or Spanish, child two or more grade levels delayed in school for reading and writing in his/her native language

Unable to read, understand or complete informed consent in English or Spanish

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Robinson, MD, MPH, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will be based on the policy for data sharing issued by the NIH and consistent with HIPAA privacy standards. Our data management team will prepare de-identified public use data set from this study for deposition in a repository.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Limited access data will be shared within six months of the publication date for the primary outcome publication or within two years of the date that the database is locked for analysis, whichever occurs first.
Access Criteria: User registration will be required. Users must agree to the conditions of use governing access to the public release data (a data use agreement), including restrictions against attempting to identify study participants, destruction of the data after analyses are completed, reporting responsibilities, restrictions on redistribution of the data to third parties, and proper acknowledgement of the data resource.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: To enter the study, the child and at least one parent/guardian must have agreed to participate, and both child and adult were considered to be enrolled.
Groups:
- Wise Interventions Plus Behavioral Rx: Participants receive Wise social psychological interventions (growth mindset and values self-affirmation) plus a 6-month usual care behavioral intervention for weight control.
- Education Plus Behavioral Rx: Participants receive health education plus a 6-month usual care behavioral intervention for weight control.
Period: Overall Study
Arm/Group | Wise Interventions Plus Behavioral Rx | Education Plus Behavioral Rx
Started | 0 | 2
Completed | 0 | 0
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Arm/Group | Education Plus Behavioral Rx
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Mass Index From Baseline to 6 Months
Description: body mass index = weight in kilograms divided by the squared height in meters
Time Frame: Change from baseline to 6 months
Population: No participant had post-baseline BMI data
Arm/Group | Education Plus Behavioral Rx
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 2.5 months, when participation ended.
Arm/Group | Education Plus Behavioral Rx
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
This study did not meet its planned enrollment and did not achieve statistical power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-04-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT04422951/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-13): https://cdn.clinicaltrials.gov/large-docs/51/NCT04422951/SAP_001.pdf